CLINICAL TRIAL: NCT02636088
Title: A Phase II Study With Oxaliplatin + 5-FU + Ceuximab and Radiotherapy for the Treatment of Non-resectable, Locally Advanced But Not Metastatic Cancer of Oesophagus or the Cardia.
Brief Title: Definitive Chemoradiotherapy and Cetuximab in the Treatment of Locally Advanced Esophageal Cancer
Acronym: LERFOX-C
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gabriella Alexandersson von Döbeln (Other)
Responsible Party: Sponsor-Investigator, Gabriella Alexandersson von Döbeln, Medical doctor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-006802-40
Record Dates: First submitted 2015-12-15; First posted 2015-12-21 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Esophageal Neoplasm
Keywords: Phase II study, clinical trial
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab (Experimental): Cetuximab is administered once a week. The initial dose is 400 mg/m2 body surface area. First Cetuximab infusion should start day 15 in cycle 1.The subsequent weekly doses are 250 mg/m2.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab

SUMMARY:
In patients with esophageal cancer, treatment with curative intent can be given to medically fit patients without distant metastases. It may consist of chemoradiotherapy or surgery alone or in combination. Surgery in combination with chemotherapy is another option. For patients who are not medically fit for surgery or with unresectable invasion in adjacent structures the only alternative with curative intent is, with current knowledge, definitive chemoradiotherapy. In the current study the investigators aim to improve prognosis for patients not suitable for surgery. Patients receive treatment with conventional chemoradiotherapy (oxaliplatin, fluorouracil and radiotherapy) with the addition of a more recently developed drug, an antibody called cetuximab.

DETAILED DESCRIPTION:
Patients are treated with three cycles of oxaliplatin and fluorouracil 750 mg/m2/24 hours, day 1-5. Each cycle lasts for 21 days. Oxaliplatin is given with 130 mg/m2 in the first cycle and in cycle 2 and 3 which are administered concomitant with radiotherapy the dose is reduced to 85 mg/m2.

A loading dose of cetuximab 400 mg/m2 is given one week before the start of radiotherapy, and thereafter 250 mg/m2 is given weekly during the course of radiotherapy.

Concomitant with chemotherapy radiotherapy to a total dose of 50 Gy is given (2 Gy once daily in 25 fractions, 5 days a week) with a photon beam linear accelerator.

After treatment patients are followed every 6 months for three years with clinical examination and a CT-scan.

ELIGIBILITY:
Inclusion Criteria:

* Histological verified squamos cell carcinoma or adenocarcinoma of the oesophagus or cardia
* Performance status WHO 0-2, age 18-75 years
* Locally advanced disease, non-resectable (T4 N0-N3 M0) or disease which is not operable for any other reason (T2/T3 N0-N3 M0)
* Adequate hematological, liver and renal function
* Written informed consent

Exclusion Criteria:

* Distant metastases
* Prior chemotherapy or radiotherapy for oesophageal cancer or cancer of the cardia
* Symptomatic peripheral neuropathy equal to or greater than NCI grade 2
* Other concomitant serious illness or medical condition that would not permit the patient to complete the study treatment or sign the informed consent
* Myocardial infarction within 6 months prior to study entry
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin) unless treated, in remission and off active treatment for greater than 2 years
* Pregnancy

Ages: 18 Years to 75 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Local tumour Control | 1 year
  Local tumour control will be measured with a computed tomography

SECONDARY OUTCOMES:
Progression-free survival | 3 years
  Tumour respons evaluation with CT-scan
Toxicity | 3 years
  Toxicity will be measured with the Common Toxicity Criteria Scale
Patterns of relapse | 3 years
  First site of recurrence will be evaluated with CT, supplemented with biopsy if indicated
Overall and disease-free survival | 3 years
  Tumour respons evaluation with CT scan
Quality of life | 3 years
  Quality of life assessed with the EORTC QLQ-C30 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella A von Döbeln, MD, Principal Investigator — Karolinska University Hospital